CLINICAL TRIAL: NCT06243367
Title: Randomized Controlled Study of Preoperative Oral Carbohydrate Loading Versus Fasting in Patients Undergoing Major Abdominal Surgery
Brief Title: Preoperative Oral Carbohydrate Loading Versus Fasting in Patients Undergoing Major Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Mohammed Taher Salem Abo-Omar, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35129/12/21
Record Dates: First submitted 2024-01-14; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Carbohydrate; Fasting; Major Abdominal Surgery
MeSH Terms: conditions — Fasting | interventions — Carbohydrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast (Control) group (Placebo Comparator): Patients were instructed to be fasting for 6 hours before surgery and received only placebo drink (200 ml clear water) two hours before surgery
  Interventions: Other: Placebo drink
- Carbohydrate group (Experimental): Patients were given a meal of cup of yogurt (100 ml) with 2 spoonful of honey (42 gm) at midnight before surgery and 200 ml of a clear carbohydrate drink on the day of surgery, 2 h before anesthesia induction. This drink consisted of 200 ml water in which two spoonful of honey were dissolved.
  Interventions: Dietary Supplement: Carbohydrate

INTERVENTIONS:
Other: Placebo drink — Patients were instructed to be fasting for 6 hours before surgery and received only placebo drink (200 ml clear water) two hours before surgery
  Arms: Fast (Control) group
Dietary Supplement: Carbohydrate — Patients were given a meal of cup of yogurt (100 ml) with 2 spoonful of honey (42 gm) at midnight before surgery and 200 ml of a clear carbohydrate drink on the day of surgery, 2 h before anesthesia induction. This drink consisted of 200 ml water in which two spoonful of honey were dissolved.
  Arms: Carbohydrate group

SUMMARY:
The aim of this study is to compare the effect of preoperative carbohydrate load versus the fasting protocol in patients undergoing major abdominal operations.

DETAILED DESCRIPTION:
The surgical patients are influenced by many stressors during operation such as the prolonged fasting hours. Importantly, these stressors are iatrogenic and have been shown to disturb homeostasis with little benefit. Surgery itself, induces an endocrine and inflammatory stress response and contributes to postoperative insulin resistance (PIR) which increased also by Preoperative fasting.

Postoperative insulin resistance is a state of reduced insulin-mediated glucose uptake in skeletal muscles and adipose tissue, with an increased glucose release due to hepatic gluconeogenesis and hyperglycemia.

Strategies to reduce the postoperative stress response and postoperative insulin resistance include shortening the preoperative fasting time via preoperative carbohydrate oral drink administration (carbohydrate load). Preoperative fasting is the first step in postoperative insulin resistance development. The traditional fasting time of 6-8 h before elective surgery to prevent pulmonary aspiration usually extends up to 12 h in anesthetic practice. Overnight fasting is a physiological state of reduced insulin sensitivity due to the normal hormonal diurnal rhythm. If patients undergo surgery in the prolonged fasted state, insulin resistance may begin even before surgery.

A preoperative carbohydrate drink acts as a morning meal, may improve insulin sensitivity and propel the patient's metabolic state towards anabolism. The rationale of this study is to compare the differences between preoperative CHO loading and a conventional fasting protocol on the postoperative insulin resistance, Glasgow prognostic score (GPS), subjective patient well-being and surgical clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 and 70 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status l & ll.
* Scheduled for elective major abdominal surgery

Exclusion Criteria:

* Disseminated malignant disease.
* Increased risk for gastric content aspiration.
* Body Mass Index (BMI) below 20 or above 30 kg/m2.
* Nutritional risk screening 2002 score above 3.
* Emergency surgery, diabetic patients, immunomodulatory therapy.
* Refusal of the patient.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
The metabolic response | 5 days postoperatively
  The patient was also subjected to further assessment by bioelectrical impedence analysis for measuring of the basal body muscle mass preoperatively and 5 days postoperatively.

SECONDARY OUTCOMES:
The postoperative inflammatory response | First day postoperative
  Postoperative inflammatory response was assessed at 6 o'clock A.M on the day of surgery (T1, basal value), 6 h after surgery (T2), at 6 o'clock A.M on postoperative day 1 (T3) .
Complications | 24 hours postoperatively
  Complications such as nausea and vomiting were assessed preoperatively and at intervals 4, 8, 12, and 24 hours postoperatively
Time of independent ambulation | 27 days postoperatively
  Time of independent ambulation will be recorded.
Postoperative discharge day | 27 days postoperatively
  Postoperative discharge day will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.